CLINICAL TRIAL: NCT05732428
Title: A PHASE 1, OPEN LABEL STUDY EVALUATING THE PHARMACOKINETICS, SAFETY, AND TOLERABILITY OF ARV-471 (PF-07850327) AS A SINGLE AGENT IN CHINESE PARTICIPANTS WITH ER+/HER2- ADVANCED BREAST CANCER
Brief Title: A Study to Learn About the Study Medicine Called Vepdegestrant (ARV-471, PF-07850327) in People With ER+/HER2- Advanced Breast Cancer in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4891018; NCT05732428 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-01-17; First posted 2023-02-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARV-471 (Experimental)
  Interventions: Drug: ARV-471

INTERVENTIONS:
Drug: ARV-471 — ARV-471 will be administered orally once daily with food (eg, a light meal of approximately 400 to 600 calories which includes a mixture of fat carbohydrates, and protein) at RP3D for monotherapy defined in study ARV-471-mBC-101, in continuous dosing over 28-day cycles

SUMMARY:
The purpose of this clinical trial is to learn about the pharmacokinetics. safety and tolerability of the study medicine (called ARV-471) for the potential treatment of advanced estrogen receptor postive and human epidermal growth factor receptor 2 negative breast cancer.

This study is seeking participants have

* ER+/HER2- advanced breast cancer
* received at least 1 line of endocrine therapy with or without CDK4/6 inhibitor
* received up to 2 prior regimens of chemotherapy for advanced setting. All participants in this study will receive ARV-471. ARV-471 will be given by mouth at home once a day. The experiences of people receiving the study medicine will be examined. This will help determine if the study medicine is safe and effective.

Participants will take part in this study until their cancer is no longer responding. During this time, they will have visits at the study clinic about every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of breast cancer with evidence of ER+/HER2- locally advanced or metastatic disease, which is not amenable to surgical resection or radiation therapy with curative intent.
* Received at least 1 line of SOC of endocrine therapy with or without CDK4/6 inhibitor for locally advanced or metastatic disease.
* Up to 2 prior regimens of chemotherapy for advanced or metastatic disease setting are allowed.

Exclusion Criteria:

* Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Participants with a history of CNS metastases or cord compression are eligible if they have been definitively treated (eg, radiotherapy, stereotactic surgery) and clinically stable (including patients with residual CNS symptoms/deficits) off enzyme-inducing anticonvulsants and steroids for at least 28 days prior to first dose of study drug.
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association Class III or IV), cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism or other clinically significant episode of thromboembolic disease, congenital long QT syndrome, Torsade de Pointes, serious conduction system abnormalities (eg, bifascicular block defined as right bundle branch and left anterior or posterior hemiblock, 3rd degree AV block), clinically important arrhythmias, left anterior hemiblock (bifascicular block), ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, atrial fibrillation of any grade.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Single dose Cmax (Maximum plasma concentration) | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose up to Day 2
  Maximum plasma concentration
Single dose AUCtau | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 2
  Area under the concentration-time profile from time zero to time tau (τ), the dosing interval, where tau = 24 hours (QD dosing)
Multiple dose Cmax | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
  Maximum Observed Plasma Concentration (Cmax)
Multiple dose AUCtau | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
  Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 24 hours.

SECONDARY OUTCOMES:
Objective Response Rate - Percentage of Participants With Objective Response | Baseline up to 24 weeks
  Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response.
  Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of Percentage of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST).
Percentage of Participants With Clinical Benefit | Baseline up to 24 weeks
  Percent of participants with confirmed complete response (CR), partial response (PR) or stable disease (SD) for at least 24 weeks on study according to RECIST.
  Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. SD was defined as not qualifying for CR, PR, Progressive Disease (PD).
Duration of Objective Response (DOR) | From the date of first documented response (CR or PR) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 weeks
  DOR: time from date of first documented response (CR or PR) to first documented progression or death due to underlying cancer. RECIST V1.1, a) CR: disappearance of all lesions; any pathological lymph nodes (TLs) or non-pathological (non-TLs) must have reduction in short axis to <10 mm; normalization of tumor marker level for non-TLs; b) PR: >=30% decrease in sum of diameter (dia) of all TLs, referring baseline sum of dia; c) PD: >=20% increase in sum of diameter of all measured target lesions taking as reference smallest sum of diameter of all target lesions recorded at or after baseline, sum must also be absolute increase of >=5 mm. Unequivocal progression of existing non-target lesions. Appearance of at least 1 new lesion. If a participant with a CR or PR had no PD or death due to underlying cancer, participants was censored at date of last adequate tumor assessment.
Presence (rate) or absence of blood biomarkers | immediately after the end of treatment
  To identify biomarkers (ESR1 mutation) of complete response and progression if occurs
Number of Participants With Notable Electrocardiogram (ECG) Values | From baseline up to 28 days after last dose of study drug
  Criteria for notable ECG values were as follow: QT interval (in millisecond [msec]) new (newly occurring post-baseline value) greater than (>) 450, 480, 500, increase from baseline >30, increase from baseline >60; corrected QT interval by Fredericia formula (QTcF) in msec new (newly occurring post-baseline value) > 450, 480, 500, increase from baseline >30, increase from baseline >60; corrected QT interval by Bazett's formula (QTcB) in msec new (newly occurring post-baseline value) > 450, 480, 500, increase from baseline >30, increase from baseline >60; heart rate in bpm new (newly occurring post-baseline value) <60 and >100.
Number of Participants With Laboratory Abnormalities | Baseline (Day 1) up to at least 28 days after last dose of study drug
  Hemoglobin (HGB),hematocrit,erythrocytes (ery.),HDL cholesterol (chl.)<0.8*lower limit of normal(LLN);reticulocytes (ret.), ret./ery. (%)<0.5*LLN,>1.5*upper limit of normal (ULN);ery. mean corpuscular (EMC) volume,EMC HGB,EMC HGB
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 28 days after last dose of study drug
  Vital signs (temperature, respiratory rate, pulse, systolic and diastolic blood pressure) were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs was determined at the investigator's discretion.
Number of Participants With Adverse Events (AEs) by type, frequency, severity (as graded by NCI CTCAE verision 5.0), timing, seriousness and relationship to study treatment | Baseline up to 28 days after the last dose of study drug
  Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] was assessed by the investigator. Participants with multiple occurrences of an AE within a category were counted once within the category. An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per CTCAE version 4, Grade 1= mild AE; Grade 2= moderate AE; Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE.
Single dose Tmax | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 2
  Time at which Cmax occurred
Single dose AUClast | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 2
  Area under the concentration-time profile from time zero to the time of the last quantifiable concentration (Clast)
Single dose MRCmax | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 2
  ARV-473 to ARV-471 ratio for Cmax
Single dose AUCinf | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 2
  Area under the concentration-time profile from time zero extrapolated to infinite time
Single dose CL/F | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 2
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Single dose Vz/F | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 2
  Apparent volume of distribution
Single dose t½ | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 2
  Terminal half-life
Multiple dose Tmax | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
  Time to Reach Maximum Observed Plasma Concentration
Multiple dose Vz/F | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
Multiple dose MRCmax | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
  ARV-473 to ARV-471 ratio for Cmax
Rac | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
  Accumulation ratio based on AUC (observed)
t½eff | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
  Effective half-life (t½eff) based on accumulation ratio
Multiple dose CL/F | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Multiple dose t½ | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
  Terminal half-life
Single dose MRAUCtau | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 2
Multiple dose AUClast | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
Multiple dose Cmin | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71
Multiple dose Ctrough | 0, 1, 2, 4, 6, 8, 12, 24 hours post-dose Up to Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Jilin Province Tumor Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891018